CLINICAL TRIAL: NCT01845610
Title: Randomized Controlled Trial in South Africa Comparing the Efficacy of Complementary Food Products on Child Growth
Acronym: TSWAKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North-West University, South Africa (Other)
Collaborators: Global Alliance for Improved Nutrition (Other); DSM Ltd (Industry); Unilever R&D (Industry)
Responsible Party: Principal Investigator, Marius Smuts, Professor, North-West University, South Africa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSWAKA
Record Dates: First submitted 2012-11-30; First posted 2013-05-03 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Fatty Acids, Essential; 6-Phytase; Lysine; Potassium; Phosphorus, Dietary; Magnesium; Manganese

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fortified fat-based paste with EFAs, DHA, ARA and phytase (Experimental): Complementary food supplement providing micronutrients and both essential fatty acids, DHA, ARA, phytase and L-lysine, potassium, phosphorous, magnesium and manganese
  Interventions: Dietary Supplement: Fortified fat-based paste with essential fatty acids, DHA, ARA, phytase, L-lysine, potassium, phosphorous, magnesium and manganese
- Fortified fat-based paste with essential fatty acids (Experimental): Complementary food supplement providing micronutrients and essential fatty acids (EFAs)
  Interventions: Dietary Supplement: Fortified fat-based paste with essential fatty acids
- Control group (No Intervention): The control group will receive a delayed intervention

INTERVENTIONS:
Dietary Supplement: Fortified fat-based paste with essential fatty acids, DHA, ARA, phytase, L-lysine, potassium, phosphorous, magnesium and manganese — Complementary food supplement providing micronutrients, essential fatty acids, DHA and ARA, phytase, L-lysine, potassium, phosphorous, magnesium and manganese
  Arms: Fortified fat-based paste with EFAs, DHA, ARA and phytase
Dietary Supplement: Fortified fat-based paste with essential fatty acids — Complementary food supplement fortified with micronutrients and essential fatty acids
  Arms: Fortified fat-based paste with essential fatty acids

SUMMARY:
Complementary food supplements (CFS), fortified products that are mixed with the infant's usual complementary foods, have the potential to improve nutrition among infants. In Africa, maize is a major staple food used for complementary feeding. Compared to rice or wheat, maize has higher levels of phytates, which bind trace elements such as iron and zinc, and inhibit their absorption. The impact of CFS products in the context of a maize-based diet has not been well investigated. This study will test two newly developed fat-based CFS products made from soy.

The first product is a fortified fat-based spread that contains essential fatty acids with added docosahexaenoic acid (DHA) and arachidonic acid (ARA), and phytase to improve iron and zinc bioavailability. The second product is a fortified fat-based product containing essential fatty acids. Both products contain soy. The enrichment of the products with essential fatty acids is of particular interest in the South African context, as consumers are exposed to higher linoleic acid (LA) diets due to the inclusion of mostly high LA-containing sunflower oil during food preparation. The CFS products could contribute towards restoring the balance between LA and alpha-linolenic acid (ALA) intake.

The results of this study will provide evidence on whether or not two types of fortified CFS have the potential to address malnutrition (linear growth) and improve psychomotor development in infants. If proven effective, this approach of providing multiple nutrients can be made available to infants in the developing world and may lead to sustainable actions.

ELIGIBILITY:
Inclusion Criteria:

* Infants resident in the study area
* Aged 6 months

Exclusion Criteria:

* Severe obvious congenital abnormalities
* Severe anaemia (haemoglobin < 70 g/L)
* Severe malnutrition (weight-for-length Z-score <-3.00)
* Other diseases referred for hospitalization by clinic staff
* Plans to move out of the study area in the next 7 months
* Known food allergies/intolerances e.g. to peanuts, milk and fish
* Infants given special nutritional supplements
* Infants known to be HIV+
* Not been borne as a singleton

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Linear growth by measuring length | 6 months
  To assess the effects of two different fortified fat-based complementary food supplements on linear growth compared to a control

SECONDARY OUTCOMES:
Psychomotor-motor development measured by the Kilifi Developmental Inventory and Parent rating (gross motor skills) at baseline and end. Motor milestones chart (weekly) | 6 months
  To investigate the effects of two different fortified fat-based complementary food supplements on psycho-motor development of infants compared to a control group.
Measures of anemia, essential fatty acid, iron and iodine status | 6 months
  To investigate the effects of two different fortified fat-based complementary food supplements on anemia, essential fatty acid, iron and iodine status of infants compared to a control group.
Growth by measuring weight of infant (bi-monthly, mid-upper arm circumference (MUAC) and head circumference of infant (baseline and end) | 6 month
  To assess the effects of two different fortified fat-based complementary food supplements on weight, MUAC and head circumference of infants

OTHER OUTCOMES:
Safety | 6 months
  Safety will be assessed by recording (serious) adverse events [(S)AEs]. This is comprised in the Record Morbidity activity. Episodes of vomit, diarrheal, upper respiratory diseases, fever and rush will be weekly monitoring and recording. A morbidity questionnaire has been purposely developed.
Nutritional status of mothers/caregivers | 6 months
  Mothers/caregivers height and weight, and a breast milk and urine sample of mothers will be taken at baseline as a reflection of their nutritional status.
Acceptability | 1 month
  Acceptability of complementary food supplements will be assessed before the start of the intervention trial
Dietary assessment | 6 months
  Multiple pass 24-hr recall (baseline and end)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius M Smuts, PhD, Principal Investigator — North-West University, South Africa
Locations (1):
- Jouberton area of the greater Matlosana Municipality, Jouberton, North West, South Africa

REFERENCES:
- [Derived] Smuts CM, Matsungo TM, Malan L, Kruger HS, Rothman M, Kvalsvig JD, Covic N, Joosten K, Osendarp SJM, Bruins MJ, Frenken LGJ, Lombard CJ, Faber M. Effect of small-quantity lipid-based nutrient supplements on growth, psychomotor development, iron status, and morbidity among 6- to 12-mo-old infants in South Africa: a randomized controlled trial. Am J Clin Nutr. 2019 Jan 1;109(1):55-68. doi: 10.1093/ajcn/nqy282. PMID 30649163